CLINICAL TRIAL: NCT02428569
Title: Providing Resources to Enhance Patients' Readiness to Make Decisions About Kidney Disease: Partnering to Break the News, Review All Options, Weigh Pros and Cons (PREPARE NOW)
Brief Title: Providing Resources to Enhance Patients' Readiness to Make Decisions About Kidney Disease: The PREPARE NOW Study
Acronym: PREPARE NOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00051812; 1R34DK094116-01 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-04-29 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Chronic Kidney Disease
Keywords: shared decision making; patient education; decision aids
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Participants randomized to this arm of the study will receive usual care from their physician.
- PREPARED Decision Support (Experimental): Participants randomized to this arm of the study will receive the PREPARED educational book and video.
  Interventions: Behavioral: PREPARED Decision Support

INTERVENTIONS:
Behavioral: PREPARED Decision Support — The PREPARED DVD presents patient and health care provider testimonials that characterize the pros and cons of different kidney replacement treatment options, including in-center hemodialysis, home hemodialysis, peritoneal dialysis, kidney transplant, and conservative management (i.e., no dialysis or transplant). The PREPARED book reinforces differences between the treatments by showing (in lay language) summaries of scientific evidence on treatment outcomes associated with each kidney replacement option.
  Arms: PREPARED Decision Support

SUMMARY:
This study evaluates the effectiveness of patient educational materials (a book and DVD) to help patients with chronic kidney disease make early, shared, and informed decisions about kidney replacement therapy. Half of the participants will receive the educational materials and half will receive usual care from their doctors.

DETAILED DESCRIPTION:
The investigators will study the effectiveness of patient educational materials (a book and DVD, called the PREPARED materials) to help patients with chronic kidney disease make early, shared, and informed decisions about kidney replacement therapy. Half of the participants will receive the PREPARED materials and half will receive usual care from their doctors. PREPARED materials feature patients and their families discussing the pros and cons of different treatment options for kidney failure. The investigators will randomly assign patients already under the care of a nephrologist to receive the video and book or to receive their usual nephrology care. They will measure the degree to which patients in either study arm are prepared for kidney failure treatment at follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Advanced kidney disease defined as an eGFR < 20 mL/min/1.73m2 at their last clinical appointment with their nephrologist
* Have not initiated a Renal Replacement Therapy

Exclusion Criteria:

* Cannot speak English
* Have initiated Renal Replacement Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Initiation of self-care dialysis or receipt of transplant | 90 days after randomization
  Among the participants initiating renal replacement therapy (RRT) during follow up, the proportion who initiate self-care dialysis (peritoneal dialysis or home hemodialysis) or receive a transplant.
Use of permanent vascular access | 90 days after randomization
  Proportion of patients achieving initiation of RRT with a permanent vascular access.
Emergent dialysis initiation | 90 days after randomization
  Proportion of patients initiating dialysis urgently in the Emergency Room (versus planned initiation).
Transplant evaluations, waiting list placement | 90 days after randomization
  Proportion of patients achieving receipt of transplant evaluations, or placement on the kidney transplant waiting list prior to initiation.
Blood pressure control at RRT initiation | 90 days after randomization
  Proportion of patients achieving blood pressure control (systolic blood pressure <130mmHg and diastolic blood pressure <80mmHg) at each visit prior to RRT initiation or completion of study follow up.
Anemia management | 90 days after randomization
  Proportion of patients with anemia treated to recommended levels (hemoglobin 10g/dl to 12g/dl) at each visit prior to RRT initiation or completion of study follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh E. Boulware, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Johns Hopkins University / Nephrology Center Of Maryland / Good Samaritan Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] DePasquale N, Ephraim PL, Ameling J, Lewis-Boyer L, Crews DC, Greer RC, Rabb H, Powe NR, Jaar BG, Gimenez L, Auguste P, Jenckes M, Boulware LE. Selecting renal replacement therapies: what do African American and non-African American patients and their families think others should know? A mixed methods study. BMC Nephrol. 2013 Jan 14;14:9. doi: 10.1186/1471-2369-14-9. PMID 23317336
- [Background] Ameling JM, Auguste P, Ephraim PL, Lewis-Boyer L, DePasquale N, Greer RC, Crews DC, Powe NR, Rabb H, Boulware LE. Development of a decision aid to inform patients' and families' renal replacement therapy selection decisions. BMC Med Inform Decis Mak. 2012 Dec 1;12:140. doi: 10.1186/1472-6947-12-140. PMID 23198793
- [Background] Sheu J, Ephraim PL, Powe NR, Rabb H, Senga M, Evans KE, Jaar BG, Crews DC, Greer RC, Boulware LE. African American and non-African American patients' and families' decision making about renal replacement therapies. Qual Health Res. 2012 Jul;22(7):997-1006. doi: 10.1177/1049732312443427. PMID 22645225